CLINICAL TRIAL: NCT01733966
Title: A Third Phase, Multicentre, Randomized as a Double Blind Study, Triple Placebo, Comparative of the Efficacy and Safety of an Association Secnidazol-Ciprofloxacin Compared With Amoxicillin-Clavulanic Acid for the Treatment of Uncomplicated Episode of Diverticular Sigmoïditis Among Adults
Brief Title: A Multicentre, Randomized as a Double Blind Study, Triple Placebo, Comparative of the Efficacy and Safety of an Association Secnidazol-Ciprofloxacin Compared With Amoxicillin-Clavulanic Acid for the Treatment of Uncomplicated Episode of Diverticular Sigmoïditis Among Adults
Acronym: DIVA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulties to recruit patients who suffer from this pathology
Sponsor: Quanta Medical (Industry)
Collaborators: Laboratoires Iprad-Vegebom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPR_SIGMO_09; NCT01136434 (obsolete NCT alias)
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2010-03

CONDITIONS: Diverticular Sigmoïditis
MeSH Terms: interventions — secnidazole; Ciprofloxacin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Secnidazol-Ciprofloxacin (Experimental): 2g(single dose) of Secnidazol associated with 1g(2 doses of 500mg)of Ciprofloxacin during 3 days
  Interventions: Drug: Secnidazole, ciprofloxacine
- Amoxicillin-Clavulanic Acid (Active Comparator): 3g (3 doses of 1g) of Amoxicillin-Clavulanic acid during 10 days
  Interventions: Drug: Amoxicillin-Clavulanic Acid

INTERVENTIONS:
Drug: Secnidazole, ciprofloxacine — 2g of microgranules of secnidazole. a single dose per day during 3 days.
  1g of Ciprofloxacin (2 tablets of 500mg per day during 3 days)
  Arms: Secnidazol-Ciprofloxacin
Drug: Amoxicillin-Clavulanic Acid — 3g of Amoxicillin-Clavulanic acid (3 powder packet of 1g per day during 10 days)
  Arms: Amoxicillin-Clavulanic Acid

SUMMARY:
The primary outcome measure is to compare efficacy of an association of Secnidazol(2g)-Ciprofloxacin(1g) (during 3 days) versus 3g of Amoxicillin-Clavulanic Acid during 10 days for the Treatment of Uncomplicated Episode of Diverticular Sigmoïditis Among Adults in clinical and biological cure.

The cure rate will be evaluated at the second visit (14 days after the inclusion visit)

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Recovering of written and dated informed consent form
* Social Security medical cover
* Left Iliac Fossa (LIF) pain
* Moderate fever (>37.8°C)
* Sensitivity/defence during LIF palpation

Biological results :

* CRP > 10mg/L
* NFS > 10G/L
* Neutrophil Granulocytosis > 75%
* Radiological results - presence to the scan :diverticul & pericolic infiltration

Exclusion Criteria:

* Patients treated by antibiotherapy in the last 15 days prior inclusion
* Patients treated by morphinic drug
* Patients treated by anticoagulant drug
* Pregnant or breast-feeding women
* Patients presenting allergy to active principal, to galactose
* Patients having taking part in another study in the last 3 months prior inclusion
* Patients unable to comply with the study requirements
* Patients presenting Chronic affection inconsistent with the study
* Patients presenting high fever
* Patients presenting abdominal contracture
* Patients presenting immunosuppression
* Radiological sign of complication (abscess>3cm)
* Patients presenting Pathology inconsistent with efficacy evaluatio

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
comparaison of the efficacy of an association of Secnidazol(2g)-Ciprofloxacin(1g) (during 3 days) versus 3g of Amoxicillin-Clavulanic Acid during 10 days for clinical and biological cure | the cure rate will be evaluated at the second visit (14 days after the inclusion visit)